CLINICAL TRIAL: NCT01101412
Title: Multi-Center, Prospective, Randomized, Double-Blinded, Controlled Clinical Trial to Evaluate the Safety and Effectiveness of an Antimicrobial Catheter Lock Solution in Maintaining Catheter Patency and Preventing Catheter Related Blood Stream Infections (CRBSI)
Brief Title: Antimicrobial Solution or Saline Solution in Maintaining Catheter Patency and Preventing Catheter-Related Blood Infections in Patients With Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was not opened.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2009-0237; MDA-2009-0237; CDR0000668850 (Other: NCI PDQ)
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Myeloproliferative Disorders; Infection; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: infection; unspecified adult solid tumor, protocol specific; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage 0 chronic lymphocytic leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated hairy cell leukemia; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders; Infections; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis | interventions — Pentetic Acid; Edetic Acid; Ethanol; ethanolamine oleate; Trimethoprim, Sulfamethoxazole Drug Combination; Trimethoprim; Sulfamethoxazole; Saline Solution, Hypertonic; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Antimicrobial Solution (Experimental): Antimicrobial solution into central or peripheral venous catheter (CVC or PVC) once daily for 90 days. Catheter dwell time is 1-24 hours. The catheter is then flushed through before any drug infusion or blood aspiration.
  Interventions: Drug: Edetate Calcium Disodium; Drug: Ethanol; Drug: Trimethoprim-sulfamethoxazole
- Arm II: Saline Solution (Active Comparator): Saline solution into CVC or PVC once daily for 90 days. Catheter dwell time is 1-24 hours. The catheter is then flushed through before any drug infusion or blood aspiration.
  Interventions: Other: Hypertonic Saline

INTERVENTIONS:
Drug: Edetate Calcium Disodium — Given through CVC or PVC.
  Other Names: Calcium Disodium Versenate; Calcium EDTA
  Arms: Arm I: Antimicrobial Solution
Drug: Ethanol — Given through CVC or PVC
  Other Names: Ethyl Alcohol; Ehtyol; Ethamolin
  Arms: Arm I: Antimicrobial Solution
Drug: Trimethoprim-sulfamethoxazole — Given through CVC or PVC
  Other Names: Bactrim; Trimethoprim; sulfamethoxazole; Bactrim DS; Cotrim DS; Septra; Sulfatrim DS; Trisulfam; Uroplus DS; Uroplus SS; Co-trimoxazole; SMX-TMP; TMP-SMX
  Arms: Arm I: Antimicrobial Solution
Other: Hypertonic Saline — Given through CVC or PVC
  Other Names: Saline; Saline Solution
  Arms: Arm II: Saline Solution

SUMMARY:
RATIONALE: Antimicrobial solution comprising trimethoprim-sulfamethoxazole, edetate calcium disodium, and ethanol may help prevent blockages and infections from forming in patients with central venous access catheters or peripheral venous catheters.

PURPOSE: This randomized trial is studying an antimicrobial solution or saline solution in maintaining catheter patency and preventing catheter-related blood infections in patients with malignancies.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the safety of antimicrobial catheter lock solution comprising trimethoprim-sulfamethoxazole, edetate calcium disodium (EDTA), and ethanol versus saline solution in patients with malignancies.
* To compare the efficacy of this lock solution versus saline solution in maintaining catheter patency in these patients.
* To demonstrate the superiority of this lock solution in preventing or reducing the incidence of catheter-related bloodstream infections in patients with long-term indwelling catheters.

OUTLINE: This is a multicenter study. Patients are stratified according to clinical site and randomized to 1 of 2 intervention arms.

* Arm I: Patients receive antimicrobial solution into the central or peripheral venous catheter (CVC or PVC) once daily for 90 days. Catheter dwell time is 1-24 hours. The catheter is then flushed through before any drug infusion or blood aspiration.
* Arm II: Patients receive saline solution into the CVC or PVC once daily for 90 days. Catheter dwell time is 1-24 hours. The catheter is then flushed through before any drug infusion or blood aspiration.

After completion of study, patients are followed up at 10 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a malignancy
* Indwelling catheter (central or peripheral) with external lumen(s) that has been in place for ≤ 7 days

  * Inpatients must have each lumen of the catheter able to be locked with the study solution uninterruptedly for a minimum of one hour per day
  * Outpatients must agree to flush and relock the catheter each day

PATIENT CHARACTERISTICS:

* Willing and able to follow the instructions required to complete the study
* No local or systemic infection as defined by the evidence of fever (e.g., body temperature ≥ 38.0 degrees C) within 24 hours including any of the following:

  * White Blood Count (WBC) ≥ 12,000/mm³ or ≤ 4,000/mm³ OR with a differential count showing ≥ 10% bands
  * Tachycardia defined as pulse rate ≥ 100 bpm
  * Tachypnea defined as respiratory rate > 20 breaths/minute
  * Hypotension defined as systolic blood pressure (BP) ≤ 90 mm Hg
  * Signs and symptoms of localized catheter-related infection (e.g., tenderness and/or pain, erythema, swelling, or purulent exudate within 2 cm of entry site)
* No occluded (partially or totally) catheter defined as inability to either withdraw blood or instill 3 cc of fluid without resistance through any catheter lumen
* No known alcohol dehydrogenase deficiency
* No known history of allergic reaction to ethanol, trimethoprim (including trimethoprim/sulfamethoxazole), or any other components within the lock solution formulation
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No renal failure or creatinine level ≥ 2.0 mg/dL
* No known heart failure or ejection fraction ≤ 25%
* No alcohol dependency

PRIOR CONCURRENT THERAPY:

* Concurrent investigational chemotherapy agents allowed

  * No concurrent non-chemotherapy investigational protocols
* Not requiring multiple central venous catheters

  * Multiple lumens in a single catheter allowed
* No catheter coated or impregnated with heparin or antimicrobial or antiseptic agent
* No concurrent routine treatment of the underlying disease that will interfere with the lock solution
* No concurrent disulfiram or metronidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence of occlusion as defined by the inability to infuse or withdraw 3 cc of saline from the catheter | 60 days
Time to development of a catheter-related bloodstream infections during the period of lock therapy administration | 60 days
Adverse events | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Chaftari, MD, Study Chair — M.D. Anderson Cancer Center; Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org